CLINICAL TRIAL: NCT00360334
Title: An Open Label Study Comparing Exenatide With Basal Insulin in Achieving an HbA1c of ≤ 7.4% With Minimum Weight Gain, in Type 2 Diabetes Patients Who Are Not Achieving Adequate HbA1c Control on Oral Anti Diabetic Therapies Alone
Brief Title: A Study Comparing Exenatide With Basal Insulin in Achieving a Target HbA1c With Minimum Weight Gain in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-BP-GWBG
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Results first posted 2009-06-05 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; exenatide; insulin glargine; Lilly; Amylin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: exenatide
- 2 (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day
  Other Names: Byetta
  Arms: 1
Drug: insulin glargine — subcutaneous injection, titrated to target blood glucose level, once a day
  Other Names: Lantus
  Arms: 2

SUMMARY:
This is a phase 3 trial designed to compare the effects of twice daily exenatide plus oral antidiabetic agents (OADs) and once-daily insulin glargine plus OADs with respect to glycemic control, as measured by hemoglobin A1c, with minimum weight gain, in patients with uncontrolled type 2 diabetes on OADs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Currently being treated with the following: Dual or triple oral therapy - on a stable combination and dose for at least 3 months.
* HbA1c between 7.5% and 10.0%.
* BMI >27.

Exclusion Criteria:

* Receive chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks immediately prior to study.
* Have participated in an interventional medical, surgical, or pharmaceutical study (a study in which a medical or surgical treatment was given) within 30 days prior to entry into the study.
* Treatment with the following medications: *Insulin as outpatient therapy within last 3 months; *Meglitinides, or acarbose within the last 3 months; *Regular use of any drugs that directly affect gastrointestinal motility; *Any previous (study) therapy with exenatide or glucagon-like peptide-1 (GLP-1) analogue; *Anti-obesity agent use within the last 3 months.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Silva de Lima, MD, Study Director — Eli Lilly and Company
Locations (31):
- United Kingdom (31):
  - Research Site, Aberdeen
  - Research Site, Bath
  - Research Site, Blackburn
  - Research Site, Bolton
  - Research Site, Bournemouth
  - Research Site, Bristol
  - Research Site, Chippenham
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Haywards Heath
  - Research Site, High Wycombe
  - Research Site, Hull
  - Research Site, Ipswich
  - Research Site, Kent
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, Livingstone
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Middlesbrough
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Oldham
  - Research Site, Oxford
  - Research Site, Plymouth
  - Research Site, Rochdale
  - Research Site, Salford
  - Research Site, Swansea
  - Research Site, Torquay
  - Research Site, Wakefield

REFERENCES:
- [Result] Davies MJ, Donnelly R, Barnett AH, Jones S, Nicolay C, Kilcoyne A. Exenatide compared with long-acting insulin to achieve glycaemic control with minimal weight gain in patients with type 2 diabetes: results of the Helping Evaluate Exenatide in patients with diabetes compared with Long-Acting insulin (HEELA) study. Diabetes Obes Metab. 2009 Dec;11(12):1153-62. doi: 10.1111/j.1463-1326.2009.01154.x. PMID 19930005
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 35 study centers in the United Kingdom. Recruitment occurred from June 2006 to October 2007.
Pre-assignment Details: One patient assigned to the Insulin Glargine group withdrew from the study prior to receiving study drug. This patient is not included in the analysis set.
Groups:
- Exenatide: 5mcg twice daily for 4 weeks, followed by 10mcg twice daily for 22 weeks
- Insulin Glargine: dosing based on treat to target protocol
Period: Overall Study
Arm/Group | Exenatide | Insulin Glargine
Started | 118 | 117
Full Analysis Set (FAS) | 118 (FAS = received ≥ 1 dose of study drug) | 116 (FAS = received ≥ 1 dose of study drug)
Completed | 99 | 104
Not Completed | 19 | 13
Not completed — Adverse Event | 7 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 2 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Entry criterion not met | 1 | 2
Not completed — Subject decision | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Insulin Glargine | Total
Number analyzed (Participants) | 118 | 116 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.2) | 56.2 (7.9) | 56.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 39 | 74
  Male | 83 | 77 | 160
Region of Enrollment [Number; unit: participants]
  United Kingdom | 118 | 116 | 234
Types of oral antidiabetic medication combinations administered at baseline [Number; unit: participants]
  metformin and sulfonylurea | 50 | 49 | 99
  metformin and thiazolidinedione | 17 | 15 | 32
  sulfonylurea and thiazolidinedione | 2 | 4 | 6
  metformin, sulfonylurea, and thiazolidinedione | 48 | 47 | 95
  other | 1 | 1 | 2
Baseline apolipoprotein-B [Mean (Standard Deviation); unit: g/L] | 0.84 (0.24) | 0.88 (0.24) | 0.86 (0.24)
Baseline fasting serum glucose [Mean (Standard Deviation); unit: mmol/L] | 10.84 (2.23) | 10.12 (2.22) | 10.48 (2.25)
Baseline fasting serum total cholesterol (TC) [Mean (Standard Deviation); unit: mmol/L] | 4.45 (1.05) | 4.63 (1.20) | 4.54 (1.13)
Baseline fasting serum triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.94 (1.01) | 2.31 (2.24) | 2.13 (1.75)
Baseline high density lipoprotein (HDL) cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.14 (0.24) | 1.15 (0.29) | 1.15 (0.27)
Baseline low density lipoprotein (LDL) cholesterol [Mean (Standard Deviation); unit: mmol/L] | 2.38 (0.82) | 2.49 (1.02) | 2.43 (0.93)
Baseline total cholesterol to high density lipoprotein cholesterol ratio [Mean (Standard Deviation); unit: ratio] | 4.00 (1.10) | 4.29 (2.15) | 4.15 (1.72)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Achieved HbA1c ≤ 7.4% With Minimal Weight Gain (≤ 1kg)
Description: Composite endpoint evaluating effect of treatment on glycemic control and weight
Time Frame: 26 weeks
Population: Full Analysis Set; The last post-baseline measurement set of both non-missing HbA1c and weight was used as endpoint value. Patients who did not have a baseline weight measurement and/or missing post-baseline measurements for HbA1c and/or weight were included in the analysis as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 116
percentage of participants | 53.4 | 19.8
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Odds Ratio (OR) = odds of a patient in the exenatide arm achieving the primary outcome divided by the odds of a patient in the insulin glargine arm achieving the primary outcome; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.71, 95% CI [2.62 to 8.46]

2. Secondary Outcome: Percent of Patients Who Achieved HbA1c ≤ 7.4% and Weight Gain ≤ 0.5kg
Description: Composite endpoint evaluating effect of treatment on glycemic control and weight
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 116
Percentage of participants | 52.5 | 16.4
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Odds Ratio (OR) = odds of a patient in the exenatide arm achieving the secondary outcome divided by the odds of a patient in the insulin glargine arm achieving the secondary outcome; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.76, 95% CI [3.11 to 10.64]

3. Secondary Outcome: Change in Fasting Serum Glucose
Description: Change in fasting serum glucose from baseline (week 0) to endpoint (week 26)
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 103 | 101
mmol/L | -2.12 (0.25) | -3.61 (0.25)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Secondary Outcome: Percent of Patients Achieving HbA1c ≤ 7.4%
Description: Percent of patients achieving specified HbA1c target at endpoint
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward. Patients with no post-baseline HbA1c measurement are regarded as non-responders in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 116
Percentage of participants | 54.2 | 61.2
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.280, Regression, Logistic; Odds Ratio (OR) = 0.75, 95% CI [0.44 to 1.26]

5. Secondary Outcome: Percent of Patients Achieving HbA1c < 7%
Description: Percent of patients achieving specified HbA1c target at endpoint
Time Frame: 26 weeks
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 116
Percentage of participants | 34.7 | 43.1
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.191, Regression, Logistic; Odds Ratio (OR) = 0.70, 95% CI [0.42 to 1.19]

6. Secondary Outcome: Percent of Patients Achieving HbA1c < 6.5%
Description: Percent of patients achieving specified HbA1c target at endpoint
Time Frame: 26 weeks
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 116
Percentage of participants | 15.3 | 11.2
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.363, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI [0.66 to 3.07]

7. Secondary Outcome: Change in 7 Point Self Monitored Blood Glucose Profile
Description: Change from baseline to endpoint in self monitored blood glucose levels measured at 7 time points during the day
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 116
mmol/L
  Pre-breakfast: Baseline (Week 0) | 9.98 (2.11) | 9.88 (2.07)
  Pre-breakfast: Change at endpoint (Week 26) | -2.01 (2.14) | -3.99 (2.39)
  2 hrs after breakfast: Baseline (Week 0) | 13.53 (3.07) | 13.33 (2.87)
  2 hrs after breakfast: Change at endpt (Week 26) | -5.09 (3.52) | -3.95 (3.89)
  Pre-lunch: Baseline (Week 0) | 9.95 (3.24) | 9.54 (2.71)
  Pre-lunch: Change at endpoint (Week 26) | -2.21 (3.11) | -2.59 (3.27)
  2 hrs after lunch: Baseline (Week 0) | 12.07 (3.27) | 11.15 (2.59)
  2 hrs after lunch: Change at endpoint (Week 26) | -3.20 (3.30) | -2.48 (3.17)
  Pre-dinner: Baseline (Week 0) | 9.95 (2.97) | 9.37 (2.73)
  Pre-dinner: Change at endpoint (Week 26) | -2.13 (2.89) | -1.46 (4.76)
  2 hrs after dinner: Baseline (Week 0) | 12.59 (3.28) | 11.80 (2.62)
  2 hrs after dinner: Change at endpoint (Week 26) | -4.59 (3.30) | -2.06 (3.22)
  Bedtime: Baseline (Week 0) | 11.63 (3.23) | 11.24 (3.05)
  Bedtime: Change at endpoint (Week 26) | -3.56 (3.19) | -2.20 (3.47)

8. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 117 | 114
kg/m^2
  Baseline (Week 0) | 34.49 (0.49) | 33.71 (0.49)
  Change at endpoint (Week 26) | -0.95 (0.11) | 1.01 (0.11)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures

9. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline to endpoint
Time Frame: 26 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 117 | 113
cm
  Baseline (Week 0) | 112.07 (1.30) | 110.64 (1.32)
  Change at endpoint (Week 26) | -2.19 (0.54) | 1.97 (0.54)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures

10. Secondary Outcome: Change in Waist-to-hip Ratio
Description: Change in waist-to-hip ratio from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 117 | 112
Ratio
  Baseline (Week 0) | 0.99 (0.01) | 0.98 (0.01)
  Change at endpoint (Week 26) | -0.02 (0.00) | 0.01 (0.00)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures

11. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 117 | 113
kg
  Baseline (Week 0) | 101.19 (1.68) | 97.93 (1.70)
  Change at endpoint (Week 26) | -2.73 (0.31) | 2.98 (0.31)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures

12. Secondary Outcome: Percent Change in Body Weight
Description: Percent change in baseline body weight at endpoint
Time Frame: 26 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 117 | 113
Percentage | -2.8 (0.3) | 3.1 (0.3)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Repeated Measures

13. Secondary Outcome: Percent of Patients Achieving 5% Weight Loss
Description: Percent of patients who lost at least 5% of baseline body weight at endpoint
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward. For change in weight, patients should have a baseline and at least one post-baseline weight measurement. Otherwise, these patients are included as non-responders in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 116
Percentage of participants | 19.5 | 0.9
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 27.91, 95% CI [3.70 to 210.54]

14. Secondary Outcome: Percent of Patients Achieving 10% Weight Loss
Description: Percent of patients who lost at least 10% of baseline body weight at endpoint
Time Frame: 26 weeks
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 116
Percentage of participants | 4.2 | 0.0

15. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 117 | 113
mmHg
  Baseline (Week 0) | 134.0 (1.5) | 134.7 (1.5)
  Change at endpoint (Week 26) | -3.6 (1.2) | 0.6 (1.2)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.014, Mixed Model Repeated Measures

16. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 117 | 113
mmHg
  Baseline (Week 0) | 79.6 (0.8) | 79.7 (0.8)
  Change at endpoint (Week 26) | -0.8 (0.7) | 0.9 (0.7)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.100, Mixed Model Repeated Measures

17. Secondary Outcome: Change in Fasting Serum Total Cholesterol (TC)
Description: Change in TC from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 105 | 108
mmol/L | -0.36 (0.07) | -0.21 (0.07)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.125, ANCOVA

18. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol
Description: Change in HDL cholesterol from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 101 | 106
mmol/L | 0.01 (0.01) | 0.02 (0.01)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.471, ANCOVA

19. Secondary Outcome: Change in TC to HDL Cholesterol Ratio
Description: Change in TC to HDL cholesterol ratio from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 101 | 106
Ratio | -0.40 (0.10) | -0.34 (0.09)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.601, ANCOVA

20. Secondary Outcome: Change in Fasting Serum Triglycerides
Description: Change in fasting serum triglycerides from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 105 | 108
mmol/L | -0.33 (0.08) | -0.38 (0.08)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.650, ANCOVA

21. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol
Description: Change in LDL cholesterol from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 95 | 101
mmol/L | -0.25 (0.06) | -0.07 (0.05)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.017, ANCOVA

22. Secondary Outcome: Change in Apolipoprotein-B
Description: Change in apolipoprotein-B from baseline to endpoint
Time Frame: 26 weeks
Population: Full Analysis Set, Last Observation Carried Forward
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 104 | 109
g/L | -0.09 (0.02) | -0.08 (0.02)
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.667, ANCOVA

23. Secondary Outcome: Incidence of Hypoglycemic Episodes
Description: Percent of total patients in each arm experiencing hypoglycemia at any point in the 26 week study
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Number; unit: percent
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 114
percent | 50.0 | 59.6
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.139, Regression, Logistic; Odds Ratio (OR) = 0.675, 95% CI [0.401 to 1.136]

24. Secondary Outcome: Incidence of Nocturnal Hypoglycemic Episodes
Description: Percent of total patients in each arm experiencing nocturnal hypoglycemia at any point in the 26 week study
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Number; unit: percent
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 114
percent | 11.9 | 29.8
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 0.317, 95% CI [0.159 to 0.630]

25. Secondary Outcome: Incidence of Severe Hypoglycemic Episodes
Description: Percent of total patients in each arm experiencing severe hypoglycemia at any point during the 26 week study
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Number; unit: percent
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 114
percent | 4.2 | 5.3
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.716, Regression, Logistic; Odds Ratio (OR) = 0.797, 95% CI [0.235 to 2.705]

26. Secondary Outcome: Hypoglycemic Rate Per 30 Days
Description: Number of hypoglycemic episodes per patient adjusted per 30 days
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Number of episodes per 30 days
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 114
Number of episodes per 30 days | 0.069 [0.000 to 0.495] | 0.164 [0.000 to 0.686]
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.113, ANCOVA on ranks

27. Secondary Outcome: Nocturnal Hypoglycemic Rate Per 30 Days
Description: Number of nocturnal hypoglycemic episodes per patient adjusted per 30 days
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Number of episodes per 30 days
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 114
Number of episodes per 30 days | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.163]
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA on ranks

28. Secondary Outcome: Severe Hypoglycemic Rate Per 30 Days
Description: Number of severe hypoglycemic episodes per patient adjusted per 30 days
Time Frame: 26 weeks
Population: Full Analysis Set
Measure: Median (Full Range); unit: Number of episodes per 30 days
Arm/Group | Exenatide | Insulin Glargine
Number analyzed (Participants) | 118 | 114
Number of episodes per 30 days | 0.000 [0.000 to 0.989] | 0.000 [0.000 to 0.328]
Statistical Analysis 1: Comparison: Exenatide vs Insulin Glargine; Test type: Superiority or Other; p = 0.740, ANCOVA on ranks

ADVERSE EVENTS:
Arm/Group | Exenatide | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 5 | 5
Other Adverse Events (participants affected / at risk) | 105 | 94
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Exenatide | Insulin Glargine
Acute myocardial infarction (Cardiac disorders) | 1/118 (1) | 0/116 (0)
Atrioventricular block complete (Cardiac disorders) | 0/118 (0) | 1/116 (1)
Campylobacter infection (Infections and infestations) | 1/118 (1) | 0/116 (0)
Cardiac failure (Cardiac disorders) | 0/118 (0) | 1/116 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0/118 (0) | 1/116 (1)
Confusional state (Psychiatric disorders) | 1/118 (1) | 0/116 (0)
Epistaxis (Musculoskeletal and connective tissue disorders) | 0/118 (0) | 1/116 (1)
Fall (Injury, poisoning and procedural complications) | 1/118 (1) | 0/116 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1/118 (1) | 0/116 (0)
Infective exacerbation of chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 0/118 (0) | 1/116 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1/118 (1) | 0/116 (0)
Renal failure acute (Renal and urinary disorders) | 1/118 (1) | 0/116 (0)
Supraventricular tachycardia (Cardiac disorders) | 1/118 (1) | 0/116 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 0/118 (0) | 1/116 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Exenatide | Insulin Glargine
Nausea (Gastrointestinal disorders) | 57/118 | 3/116
Nasopharyngitis (Infections and infestations) | 24/118 | 23/116
Diarrhoea (Gastrointestinal disorders) | 22/118 | 14/116
Headache (Nervous system disorders) | 17/118 | 18/116
Vomiting (Gastrointestinal disorders) | 25/118 | 6/116
Lower respiratory tract infection (Infections and infestations) | 10/118 | 12/116
Abdominal distension (Gastrointestinal disorders) | 19/118 | 1/116
Dyspepsia (Gastrointestinal disorders) | 20/118 | 0/116
Early satiety (General disorders) | 20/118 | 0/116
Flatulence (Gastrointestinal disorders) | 18/118 | 1/116
Influenza (Infections and infestations) | 8/118 | 11/116
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/118 | 15/116
Arthralgia (Musculoskeletal and connective tissue disorders) | 5/118 | 12/116
Cough (Respiratory, thoracic and mediastinal disorders) | 4/118 | 13/116
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5/118 | 10/116
Back pain (Musculoskeletal and connective tissue disorders) | 5/118 | 9/116
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14/118 | 0/116
Eructation (Gastrointestinal disorders) | 13/118 | 0/116
Abdominal Pain (Gastrointestinal disorders) | 12/118 | 0/116
Anorexia (Metabolism and nutrition disorders) | 11/118 | 1/116
Dysgeusia (Nervous system disorders) | 10/118 | 0/116
Rash (Skin and subcutaneous tissue disorders) | 6/118 | 4/116
Oedema peripheral (General disorders) | 1/118 | 8/116
Injection site bruising (General disorders) | 6/118 | 2/116
Pain (General disorders) | 2/118 | 6/116
Bowel sounds abnormal (Gastrointestinal disorders) | 7/118 | 0/116
Dizziness (Nervous system disorders) | 6/118 | 1/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days